CLINICAL TRIAL: NCT07226076
Title: Reduction of Post-op Pain and Opioid Consumption With the Addition of Methadone in Total Knee Arthroplasty: a Double-blind Randomized Control Trial
Brief Title: Methadone in TKA for Post-op Pain and Opioid Reduction
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, William Barrett, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00147447
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain
Keywords: post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone (Active Comparator): Patients will intraoperatively receive methadone 0.15mg/kg IV, based on ideal body weight.
  Interventions: Drug: Methadone Hydrochloride
- No Methadone (No Intervention): Patients will NOT receive methadone.

INTERVENTIONS:
Drug: Methadone Hydrochloride — Patients will intraoperatively be administered methadone 0.15mg/kg IV, based on ideal body weight.
  Arms: Methadone

SUMMARY:
This randomized, double-blind controlled trial investigates whether intraoperative IV methadone (0.15 mg/kg based on ideal body weight) reduces acute postoperative pain and opioid consumption in patients undergoing elective total knee arthroplasty under spinal anesthesia with mepivacaine.

ELIGIBILITY:
Inclusion

* Ages 18-75 years of age
* Undergoing elective primary total knee arthroplasty with mepivacaine in the spinal anesthesia

Exclusion

* Allergy to methadone or mepivacaine
* Severe liver disease defined as Child's Pugh Class C
* End stage renal disease requiring dialysis
* Known diagnosis of prolonged QT syndrome
* Currently pregnant
* Unable to provide written, informed consent
* Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Patient reported pain in the recovery unit after surgery | up to 24 hours after surgery ends
  Patient reported pain on a Visual Analog Scale (VAS) from 0-100mm at approximately 30-60 minutes after arriving to the recovery unit after surgery. A lower pain score means a better outcome.

SECONDARY OUTCOMES:
Opioid Consumption in the recovery unit | PACU Arrival until PACU Discharge up to 30 days
  Opioid consumption measured in oral morphine milligram equivalents (MMEs) while the patient is in the PACU (Post-Anesthesia Recovery Unit).
Time to first opioid rescue dose | up to 24 hours after surgery ends
  Measured from the PACU arrival time, to the time the first opioid rescue dose is given while in the PACU.
Pain scores | PACU, 24 hours, 48 hours, and 72 hours post-operatively.
  Visual Analog Score (VAS) 0-100mm reporting pain at rest, and with movement. A lower pain score means a better outcome.
Postoperative nausea and/or vomiting | PACU through 72 hours post-operatively
  Incidence of postoperative nausea and/or vomiting after surgery as reported by the patient.
Quality of Recovery | up to 24-hours post-operatively
  Change in quality of recovery score from baseline to 24-hours post-operatively measured using the Quality of Recovery 15 Assessment (QoR-15). This assessment is scored 0-150, with a higher score indicating a better quality of recovery. Each of the 15 questions is on an 11-point numerical rating scale from 0-10, and the selections are added together to result in the total score.

CONTACTS AND LOCATIONS:
Overall Officials: William Barrett, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No